CLINICAL TRIAL: NCT03871842
Title: Study on the Safety and Effects of Transcranial Direct Current Stimulation (tDCS) in the Treatment of Depressive Symptoms in Participants With Temporal Lobe Epilepsy: A Randomized, Double-blind, Sham-controlled Clinical Trial
Brief Title: Effects of tDCS on Depressive Symptoms of Participants With Temporal Lobe Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-0352
Record Dates: First submitted 2019-02-26; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2018-07

CONDITIONS: Depressive Symptoms; Epilepsy, Temporal Lobe
MeSH Terms: conditions — Depression; Epilepsy, Temporal Lobe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS (Active Comparator): 20-minute of daily anodal stimulation (2mA) above the left dorsolateral prefrontal cortex during 5 days per week for 4 weeks.
  Interventions: Device: active tDCS
- sham tDCS (Sham Comparator): 20-minute of daily sham stimulation above the left dorsolateral prefrontal cortex during 5 days per week for 4 weeks.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: active tDCS — Considering that the daily outpatient use of tDCS equipment is not feasible for most patients, the Pain and Neuromodulation group of the Hospital de Clínicas de Porto Alegre developed a portable tDCS device for home use that has a safe protocol, in addition of being easy to use so that the patient can use it at home without help. The safety protocol embedded in the device does not, for example, allow the appliance to be used for more than 20 minutes per day. The device can also provide the assisting staff with data such as the time the patient used the equipment, providing an accurate picture of the patient's adherence to this type of equipment. This tDCS equipment for home use has already been validated in a pilot study and will be used in this work.
  Arms: active tDCS
Device: sham tDCS — The sham intervention will be applied exactly equal to active intervention, but the electric stimulus will last just for 30 seconds.
  Arms: sham tDCS

SUMMARY:
This project was developed to analyze the clinical, biochemical and functional impact of tDCS on depressive symptoms in participants with temporal lobe epilepsy, intending to collaborate directly in the development of new therapeutic strategies for participants with epilepsy and associated mood disorders. Another objective of this work is to add knowledge about biosafety, possible behavioral and electrophysiological effects of tDCS in participants with temporal lobe epilepsy. Depending on the findings, the study as proposed may provide immediate results for the care of participants with epilepsy.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) has emerged as an alternative tool in the treatment of participants with mood disorders and may also benefit the treatment of participants with epilepsy. However, this therapeutic tool has been little explored in the treatment of mood disorders in participants with epilepsy. Considering these aspects, the main objective of this project is to study the safety and possible therapeutic effects of tDCS in depressive symptoms of participants with temporal lobe epilepsy. As secondary objectives, stands out the evaluation of the effects of this stimulation on the frequency of epileptic seizures and on electrophysiological and biochemical parameters in these participants. To do this, after performing semi-structured interviews to evaluate depressive symptoms, quality of life and sleep, participants with Temporal Lobe Epilepsy will be randomized into two groups: 1) intervention with tDCS in participants with Temporal Lobe Epilepsy and depressive symptoms (T) and 2) sham intervention in participants with Temporal Lobe Epilepsy and depressive symptoms (S). After studying and characterizing the behavioral, biochemical and electroencephalic patterns (EEG), the T group will be submitted to tDCS. The control group will perform the same assessments and the same preparatory procedures, but will not receive the electrical stimulus. Finally, in addition to the analysis of the electroencephalographic patterns of the two groups at the end of each session, the analysis of the brain-derived Neurotrophic Factor Neurotrophic Factor (BDNF) will also be performed, as well as a new clinical evaluation regarding the frequency of seizures and patterns of these participants through the same semi-structured interviews conducted initially.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years.
2. Diagnosis of Temporal Lobe Epilepsy based on clinical, electrophysiological, magnetic resonance (MRI) and computed tomography (CT) imaging of the brain.
3. Patients will be selected who are able to adequately complete the self-administered questionnaires and handle the home tDCS equipment.
4. 13 points or more on the Beck Depression Inventory.

Exclusion Criteria:

1. Clinical history suggestive of other paroxysmal abnormalities other than temporal lobe epilepsy, such as syncope, psychogenic seizures, or transient vascular accident;
2. Change in the antiepileptic regime in the last 30 days;
3. History of status epilepticus on last year;
4. Performed vagus nerve stimulation (VNS), Deep Brain Stimulation (DBS) or other neurostimulation <1 year prior to study;
5. Active suicide plane;
6. Contraindication for tDCS, including head injury, metal on the head or any implanted medical device, including pacemakers and cardiac defibrillators;
7. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms, measured by Beck Depression Inventory. | 2 months
  The objective of this work is to evaluate the antidepressant effect of transcranial direct current stimulation in participants with temporal lobe epilepsy, measuring the depressive symptoms by Beck Depression Inventory before and after treatment, which score ranges from 0 to 21. High values represent more severe depressive symptoms.

SECONDARY OUTCOMES:
Seizure frequency measured by crisis diary | 3 months
  To analyze if tDCS improves the frequency of seizures observing the crisis diary during one month before and one month after treatment.
Interictal discharge counting, using Electroencephalographic Exam | 2 months
  To evaluate if epilepsy is affected by tDCS, it will be counted how many interictal discharge the participant presents before and after treatment.
Brain-Derived Neurotrophic Factor (BDNF) | 2 months
  To explore possible changes of BDNF in the groups at three times (before treatment, after 20 days of treatment and after the follow-up period), and possible correlation with the clinical findings. BDNF will be measured in Picograms Per Millilitre (pg/mL).
QOLIE-31 scale | 2 months
  To observe if there is an improvement in the quality of life of these participants, through the increase of points in the Quality of Life in Epilepsy scale (QOLIE-31), which score ranges from 0-100. High values represent better quality of life.
Pittsburgh Sleep Quality Questionnaire | 2 months
  To observe if there is improvement in sleep patterns of the participants, through Pittsburgh Sleep Quality Questionnaire, which score ranges from 0 to 21 (high scores represent better quality of sleep).
Munich Chronotype Questionnaire (MCTQ) | 2 months
  To observe if there is change in the chronotype of these participants, through Munich Chronotype Questionnaire (MCTQ).

CONTACTS AND LOCATIONS:
Overall Officials: Suelen Mota, Study Chair — HCPA
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mota SM, Amaral de Castro L, Riedel PG, Torres CM, Bragatti JA, Brondani R, Secchi TL, Sanches PRS, Caumo W, Bianchin MM. Home-Based Transcranial Direct Current Stimulation for the Treatment of Symptoms of Depression and Anxiety in Temporal Lobe Epilepsy: A Randomized, Double-Blind, Sham-Controlled Clinical Trial. Front Integr Neurosci. 2021 Dec 8;15:753995. doi: 10.3389/fnint.2021.753995. eCollection 2021. PMID 34955774